CLINICAL TRIAL: NCT03946657
Title: A Comparison of Cerebral Oximetry After Propofol-Based Total Intravenous Anesthesia and Sevoflurane Inhalation Anesthesia in Morbidly Obese Patients Undergoing LSG: a Prospective, Single-Blinded, Randomized, Parallel-Group Study.
Brief Title: Anesthetics and Cerebral Oxygenation in LSG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Cengiz KAYA, Associate Professor, MD, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: B.30.2.ODM.0.20.08/27-230
Record Dates: First submitted 2019-05-07; First posted 2019-05-10 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Morbid Obesity; Bariatric Surgery Candidate; Anesthesia
Keywords: Bariatric; Surgery; Sevoflurane; Propofol; Oximetry
MeSH Terms: conditions — Obesity, Morbid | interventions — Anesthetics, Intravenous

STUDY DESIGN:
Intervention Model Description: For the investigation, the patients were randomly assigned to two groups; the Inhalation group including those who received sevoflurane-remifentanil for the maintenance of anesthesia (n = 30) and the TIVA (total intravenous anesthesia) group including those who had propofol-remifentanil infusion for the maintenance of anesthesia (n = 30). The anesthesiologist caring for the patient was aware of the group assignments. The patients were blinded to the group assignments.
Who Masked: Participant
Masking Description: The patients were randomly assigned using opaque sealed envelopes to two groups; the Inhalation group including those who received sevoflurane-remifentanil for the maintenance of anesthesia (n = 30) and the TIVA (total intravenous anesthesia) group including those who had propofol-remifentanil infusion for the maintenance of anesthesia (n = 30). Randomization was performed according to a computer-generated randomization code, and a statement showing the patients' group was placed in sealed, numbered enveloped according to the results. Each patient drew an envelope and was enrolled in the study depending on the group written in the envelope. Randomization was performed by a physician who was not involved in the monitorization of the patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Inhalation Group (Active Comparator): Sevoflurane (1 minimum alveolar concentration [MAC]) were used in the Inhalation group for the maintenance of anesthesia.
  Interventions: Drug: Inhalational anesthetic
- The TIVA (total intravenous anesthesia) Group (Active Comparator): Propofol infusion (4-8 mg/kg of total body weight/h) were used in the TIVA group.
  Interventions: Drug: Intravenous anesthetic

INTERVENTIONS:
Drug: Inhalational anesthetic — Oxygen/air (fraction of inspired oxygen (FiO2) of 0.40), inspiratory fresh gas flow of 2 L/min), sevoflurane (1 minimum alveolar concentration [MAC]) and remifentanil IV infusion (0.1-0.25 mcg/kg of LBW/min) were used.Neuromuscular blockade was performed during the operation by rocuronium infusion (0.3-0.7 mg/kg of LBW/h), ensuring that PTC was zero.
  Arms: The Inhalation Group
Drug: Intravenous anesthetic — Propofol infusion (4-8 mg/kg of total body weight/h), oxygen/air (FiO2 of 0.40; inspiratory fresh gas flow of 2 L/min) and remifentanil IV infusion (0.1-0.25 μg/kg of LBW/min) were used.Neuromuscular blockade was performed during the operation by rocuronium infusion (0.3-0.7 mg/kg of LBW/h), ensuring that PTC was zero.
  Arms: The TIVA (total intravenous anesthesia) Group

SUMMARY:
Obesity is a global health issue that affects different organ systems and may cause severe health issues. Patients with a BMI > 40 kg/m2 or those with a BMI > 35 kg/m2 with accompanying comorbidities are candidates for weight loss surgeries, which are generally referred to as bariatric surgeries. Laparoscopic sleeve gastrectomy (LSG) is a restrictive bariatric surgery procedure gaining increased popularity in the surgical treatment of morbid obesity. However, LSG requires a reverse-Trendelenburg position and prolonged pneumoperitoneum. Carbon dioxide pneumoperitoneum increases intracranial pressure (ICP) by increasing intra-abdominal pressure and by causing dilation of cerebral vessels through carbon dioxide reabsorption. Also, the reverse-Trendelenburg position decreases cardiac output and mean arterial pressure (MAP) by reducing cardiac venous return. A Near-infrared spectroscopy (NIRS) is a non-invasive technique and provides continuous monitoring of regional cerebral tissue oxygen saturation (rSO2).

Sevoflurane and propofol are widely used for the maintenance of general anesthesia during bariatric surgery. Sevoflurane is an efficacious halogenated inhalational anesthetic for bariatric surgery because of its rapid and consistent recovery and because it does not cause hemodynamic instability because of its low blood solubility. Moreover, it increases global CBF through a direct intrinsic cerebral vasodilatory action and, in addition, it might improve cerebral oxygenation by decreasing the cerebral metabolic rate of oxygen (CMRO2) (luxury perfusion). Propofol can also be a suitable option for the maintenance of anesthesia in bariatric surgery. Propofol is a short-acting intravenous anesthetic agent with a very good recovery profile, and its elimination half-life and duration of action do not change in obese individuals. However, it has been reported that propofol may significantly decrease CBF by both suppressing CMRO2 and through a direct vasoconstrictive action. The impact of propofol on global CBF is more salient than that on CMRO2, resulting in a decrease in rSO2. The aim of the present study was to test the hypothesis that rSO2 is better preserved with sevoflurane than propofol in morbidly obese patients who have undergone LSG.

DETAILED DESCRIPTION:
All patients were administered 300 mg of oral ranitidine the night before the surgery and 10 mg intravenous (IV) metoclopramide in combination with 150 mg ranitidine one hour before arrival to the operating room. Upon the arrival to the operating room, an electrocardiogram, noninvasive blood pressure, SpO2, rSO2 (INVOSTM 5100C oximeter; Covidien, Massachusetts, USA) and neuromuscular monitorization (TOF-WatchTM SX, Organon, Dublin, Ireland) were performed on the patients. Afterwards, preoxygenation was performed with 4 L/min oxygen (80%) for three minutes by using facemasks, and anesthesia was induced with an IV propofol injection (1.5-2.5 mg/kg of ideal body weight) and an IV bolus administration of remifentanil [1 mcg/kg of lean body weight (LBW)] for 30-60 s, and then switched to infusion at 0.25 mcg/kg of LBW/min. After the eyelid reflex disappeared, a neuromuscular blockade was performed using rocuronium (1.2 mg/kg of LBW), ensuring that the train-of-four count and the post-tetanic count (PTC) were both zero, and performed tracheal intubation. Mechanical ventilation was performed with a Draeger FabiusTM Plus anesthesia workstation (Draeger Medical, Lübeck, Germany), and volume-controlled mechanical ventilation was applied. Breathing gases (oxygen, carbon dioxide, sevoflurane) were measured using Draeger ScioTM gas measurement module (Draeger Medical, Lübeck, Germany). The tidal volume was set as 7-8 mL/kg of LBW, inspiratory: expiratory ratio as 1:2, positive end-expiratory pressure as 5-8 cmH2O, and the respiratory rate was determined to obtain an end-tidal carbon dioxide partial pressure (PETCO2) of 32-37 mmHg. These ventilator settings were not changed throughout the operation. Furthermore, after the induction of anesthesia, a radial arterial line was placed in all patients for the continuous measurement of mean arterial pressure and intermittent arterial blood gas analysis.

Oxygen/air (fraction of inspired oxygen (FiO2) of 0.40), inspiratory fresh gas flow of 2 L/min), sevoflurane (1 minimum alveolar concentration [MAC]) and remifentanil IV infusion (0.1-0.25 mcg/kg of LBW/min) were used in the Inhalation group for the maintenance of anesthesia. Propofol infusion (4-8 mg/kg of total body weight/h), oxygen/air (FiO2 of 0.40; inspiratory fresh gas flow of 2 L/min) and remifentanil IV infusion (0.1-0.25 μg/kg of LBW/min) were used in the TIVA group. Neuromuscular blockade was performed during the operation by rocuronium infusion (0.3-0.7 mg/kg of LBW/h), ensuring that PTC was zero. IV normal saline or lactated Ringer's solution at 5-7 mL/kg of LBW was also used for perioperative fluid maintenance. Nasopharyngeal temperature was monitored throughout the surgery, and the patient temperature (36-37°C) was ensured by using a forced-air warming system for the maintenance of intraoperative normothermia during the procedure.

After anesthesia induction, a neutral head position of the patients was preserved to prevent alteration of cerebral venous drainage. Carbon dioxide insufflation was performed with an electronic laparoflator using a closed Veress needle technique, and intra-abdominal pressure was automatically kept at the desired level (14-16 mmHg) during the surgery. After the insufflation of carbon dioxide, the patients were positioned in a 30° reverse-Trendelenburg and at a 10° right lateral position.

At the end of the surgery, the blockade was reversed by administering 4 mg/kg of adjusted body weight sugammadex with a PTC of 1-2. All patients were extubated in the beach chair position when fully awake. The patients were referred to the recovery unit and monitored for 50 minutes for complications. In cases where no complications were apparent, the recovery was evaluated using the modified Aldrete scoring system. Once the score was ≥9, the patients were taken to unit. For postoperative nausea and vomiting, 4-5 mg dexamethasone was used (except for diabetic patients on insulin) 90 min before anesthesia induction and 4-8 mg IV ondansetron 20-30 min before the end of the operation. For postoperative pain management, 1 g IV acetaminophen was administered 20 min after induction and 30 mg IV ketorolac 20 min before onset. Then, 1 g IV acetaminophen was administered every 6 h + 50 mg IV dexketoprofen every 8 h for the first 48 hours. In addition, morphine was administered using a patient-controlled analgesia delivery system (demand dose, 20 µg/kg of ideal body weight; lockout time, 6-10 min; 4 h limit, 80% of the total calculated dosage) for 48 h postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* The American Society of Anaesthesiologists (ASA) physical status class II-III
* BMI of ≥ 35 kg/m2
* Patients were planning on undergoing an elective laparoscopic sleeve gastrectomy (LSG)

Exclusion Criteria:

* Patients with preexisting cerebrovascular diseases, overt neurological signs, alcohol or psychoactive drug addiction
* Uncontrolled diabetes or hypertension
* Advanced organ failure
* Preoperative peripheral oxygen saturation (SpO2) less than 96%
* Hemoglobin <9 g/dL .

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-01-20 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Cerebral oxygen saturation | The rSO2 values of the patients were recorded from baseline untill 20 minutes after the extubation, up to 120 min.
  The rSO2 values of the patients were recorded preoperatively, one minute after the induction, and every five minutes until the patient was referred to the recovery unit. Measurements in the last 30 seconds of preoxygenation, performed for three minutes with 4 L/min oxygen (80%) pre-induction, were accepted as preoperative values.Cerebral oxygen desaturation was defined as a greater than 25% decrease in the rSO2 value compared to the preoperative value (decrease should be more than 20% if the preoperative value is <50) and maintenance of this situation for ≥15 seconds. In this case, the following algorithm was used. First of all, normotension of the patient was ensured (administration of vasopressors such as ephedrine, and/or infusion of isotonic fluids) and the patient's neck was checked. External factors causing arterial or venous obstruction were restored, if any. If no recovery was seen despite these steps, FiO2 was set at 100%.
Arterial Blood Gas (ABG) analysis-pH | The pH values of the patients were recorded after anesthesia induction until the patient was referred to the recovery unit, up to 120 min.
  The pH values of the patients were measured in the fifth minute post-induction with the patient in the neutral position, in the 30th minute post-insufflation in the reverse-Trendelenburg position of patient and post-extubation right before the patient was referred to the recovery unit.
Arterial Blood Gas (ABG) analysis-Partial pressure of carbon dioxide | The partial pressure of carbon dioxide values of the patients were recorded after anesthesia induction until the patient was referred to the recovery unit, up to 120 min.
  The partial pressure of carbon dioxide values of the patients were measured in the fifth minute post-induction with the patient in the neutral position, in the 30th minute post-insufflation in the reverse-Trendelenburg position of patient and post-extubation right before the patient was referred to the recovery unit.
Arterial Blood Gas (ABG) analysis-Hemoglobin | The hemoglobin values of the patients were recorded after anesthesia induction until the patient was referred to the recovery unit, up to 120 min.
  The hemoglobin values of the patients were measured in the fifth minute post-induction with the patient in the neutral position, in the 30th minute post-insufflation in the reverse-Trendelenburg position of patient and post-extubation right before the patient was referred to the recovery unit.

SECONDARY OUTCOMES:
The heart rate (HR) measurement | The heart rate was recorded from baseline until the patient was referred to the recovery unit, up to 120 min.
  The heart rate was recorded preoperatively, one minute after the induction, and every five minutes until the patient was referred to the recovery unit. HR values were allowed to fluctuate up to 20% of the preoperative values of the patients. For this purpose, the infusion rate of remifentanil was accordingly increased and decreased. Whenbradycardia (HR <45 beats/minute) continued for longer than three minutes, they were treated with IV 0.5 mg atropine.
The oxygen saturation measurement | The oxygen saturation was recorded from baseline until the patient was referred to the recovery unit, up to 120 min.
  The oxygen saturation was recorded preoperatively, one minute after the induction, and every five minutes until the patient was referred to the recovery unit.
The mean arterial pressure measurement | The mean arterial pressure was recorded from baseline until the patient was referred to the recovery unit, up to 120 min.
  The mean arterial pressure was recorded preoperatively, one minute after the induction, and every five minutes until the patient was referred to the recovery unit.
The end-tidal carbon dioxide partial pressure measurement | The end-tidal carbon dioxide partial pressure was recorded from baseline until the patient was referred to the recovery unit, up to 120 min.
  The end-tidal carbon dioxide partial pressure was recorded preoperatively, one minute after the induction, and every five minutes until the patient was referred to the recovery unit.
The anesthesia time (min) | The anesthesia time was recorded through study completion.
  The anesthesia time was defined as the length of time the patient was anesthetized.
The reverse-Trendelenburg time (min) | The reverse-Trendelenburg time was recorded through study completion.
  The reverse-Trendelenburg time was defined as the length of time the patient was in the reverse-Trendelenburg position.
The pneumoperitoneum time (min) | The pneumoperitoneum time was recorded through study completion.
  The pneumoperitoneum time was defined as the length of time the patient had pneumoperitoneum
The recovery time (min) | The recovery time was recorded at the end of the surgery untill the extubation.
  The recovery time was defined as the time from discontinuation of sevoflurane or propofol and remifentanil at the end of the surgery to the restoration of spontaneous breathing, opening of the eyes upon a verbal command, squeezing of the hand of the observer and extubation.

CONTACTS AND LOCATIONS:
Overall Officials: CENGIZ KAYA, Assoc. Prof., Principal Investigator — Ondokuz Mayis University, School of Medicine, Department of Anesthesiology
Locations (1):
- Ondokuz Mayis Universitesi, Samsun, Atakum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Soleimanpour H, Safari S, Sanaie S, Nazari M, Alavian SM. Anesthetic Considerations in Patients Undergoing Bariatric Surgery: A Review Article. Anesth Pain Med. 2017 Jul 11;7(4):e57568. doi: 10.5812/aapm.57568. eCollection 2017 Aug. PMID 29430407
- [Background] Schofield DL, Morton PG, Brokos C, Gruel R, Johannes S, McBride N, et al. Perioperative Assessment and Risk Stratification of the Obese Patient. Bariat Nurs Surg Pat 2011;6:201 - 206.
- [Background] Himpens J, Dobbeleir J, Peeters G. Long-term results of laparoscopic sleeve gastrectomy for obesity. Ann Surg. 2010 Aug;252(2):319-24. doi: 10.1097/SLA.0b013e3181e90b31. PMID 20622654
- [Background] Yorulmaz IS, Demiraran Y, Salihoglu Z, Umutoglu T, Ozaydin I, Dogan S. Effect of PEEP, Zero PEEP and Intraabdominal Pressure Levels on Cerebral Oxygenation in the Morbidly Obese Undergoing Sleeve Gastrectomy. Bariatr Surg Pract P 2017;12:123 - 129.
- [Background] Willeumier KC, Taylor DV, Amen DG. Elevated BMI is associated with decreased blood flow in the prefrontal cortex using SPECT imaging in healthy adults. Obesity (Silver Spring). 2011 May;19(5):1095-7. doi: 10.1038/oby.2011.16. Epub 2011 Feb 10. PMID 21311507
- [Background] Sollazzi L, Perilli V, Modesti C, Annetta MG, Ranieri R, Tacchino RM, Proietti R. Volatile anesthesia in bariatric surgery. Obes Surg. 2001 Oct;11(5):623-6. doi: 10.1381/09608920160557138. PMID 11594107
- [Background] Kaisti KK, Langsjo JW, Aalto S, Oikonen V, Sipila H, Teras M, Hinkka S, Metsahonkala L, Scheinin H. Effects of sevoflurane, propofol, and adjunct nitrous oxide on regional cerebral blood flow, oxygen consumption, and blood volume in humans. Anesthesiology. 2003 Sep;99(3):603-13. doi: 10.1097/00000542-200309000-00015. PMID 12960544
- [Background] Servin F, Farinotti R, Haberer JP, Desmonts JM. Propofol infusion for maintenance of anesthesia in morbidly obese patients receiving nitrous oxide. A clinical and pharmacokinetic study. Anesthesiology. 1993 Apr;78(4):657-65. doi: 10.1097/00000542-199304000-00008. PMID 8466066
- [Background] Engelhard K, Werner C. Inhalational or intravenous anesthetics for craniotomies? Pro inhalational. Curr Opin Anaesthesiol. 2006 Oct;19(5):504-8. doi: 10.1097/01.aco.0000245275.76916.87. PMID 16960482
- [Background] Honca M, Honca T. Comparison of Propofol with Desflurane for Laparoscopic Sleeve Gastrectomy in Morbidly Obese patients: A Prospective Randomized Trial. Bariatr Surg Pract P 2017;12:49 - 54.
- [Background] Reinsfelt B, Westerlind A, Ricksten SE. The effects of sevoflurane on cerebral blood flow autoregulation and flow-metabolism coupling during cardiopulmonary bypass. Acta Anaesthesiol Scand. 2011 Jan;55(1):118-23. doi: 10.1111/j.1399-6576.2010.02324.x. Epub 2010 Oct 7. PMID 21039354
- [Background] Dagal A, Lam AM. Cerebral autoregulation and anesthesia. Curr Opin Anaesthesiol. 2009 Oct;22(5):547-52. doi: 10.1097/ACO.0b013e32833020be. PMID 19620861
- [Background] Klein KU, Schramm P, Glaser M, Reisch R, Tresch A, Werner C, Engelhard K. Intraoperative monitoring of cerebral microcirculation and oxygenation--a feasibility study using a novel photo-spectrometric laser-Doppler flowmetry. J Neurosurg Anesthesiol. 2010 Jan;22(1):38-45. doi: 10.1097/ANA.0b013e3181bea439. PMID 19816204
- [Background] Klein KU, Fukui K, Schramm P, Stadie A, Fischer G, Werner C, Oertel J, Engelhard K. Human cerebral microcirculation and oxygen saturation during propofol-induced reduction of bispectral index. Br J Anaesth. 2011 Nov;107(5):735-41. doi: 10.1093/bja/aer227. Epub 2011 Jul 31. PMID 21862494
- [Background] Jeong H, Jeong S, Lim HJ, Lee J, Yoo KY. Cerebral oxygen saturation measured by near-infrared spectroscopy and jugular venous bulb oxygen saturation during arthroscopic shoulder surgery in beach chair position under sevoflurane-nitrous oxide or propofol-remifentanil anesthesia. Anesthesiology. 2012 May;116(5):1047-56. doi: 10.1097/ALN.0b013e31825154d2. PMID 22421420
- [Background] Valencia L, Rodriguez-Perez A, Kuhlmorgen B, Santana RY. Does sevoflurane preserve regional cerebral oxygen saturation measured by near-infrared spectroscopy better than propofol? Ann Fr Anesth Reanim. 2014 Apr;33(4):e59-65. doi: 10.1016/j.annfar.2013.12.020. Epub 2014 Feb 24. PMID 24582111
- [Background] Ruzman T, Simurina T, Gulam D, Ruzman N, Miskulin M. Sevoflurane preserves regional cerebral oxygen saturation better than propofol: Randomized controlled trial. J Clin Anesth. 2017 Feb;36:110-117. doi: 10.1016/j.jclinane.2016.10.010. Epub 2016 Dec 1. PMID 28183546
- [Background] Sen P, Izdes S, But A. Effects of sevoflurane and propofol anaesthesia on cerebral oxygenation during normocapnia and mild hypercapnia: a pilot study. Br J Anaesth. 2013 Feb;110(2):318-9. doi: 10.1093/bja/aes489. No abstract available. PMID 23319678